CLINICAL TRIAL: NCT03968744
Title: A Prospective, Open Label, Single Arm, Clinical Study to Evaluate the Effect of Safinamide on Sleep Quality and Polysomnographic Parameters in Patients With Parkinson's Disease: the Safe Sleep Study
Brief Title: Effect of Safinamide on Sleep Quality in Patients With Parkinson's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Alain Kaelin (Other)
Collaborators: Clinical Trial Unit Ente Ospedaliero Cantonale (Other)
Responsible Party: Sponsor-Investigator, Alain Kaelin, Director of Neurocenter of Southern Switzerland, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NSI-SAF-001
Record Dates: First submitted 2019-04-19; First posted 2019-05-30 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Parkinson's Disease (at Later Stage)
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safinamide (Experimental): PO treatment: 2 weeks of treatment at dose 50 mg/day followed by 10 weeks at 100 mg/day
  Interventions: Drug: Safinamide

INTERVENTIONS:
Drug: Safinamide — Safinamide taken per Os for 12 weeks
  Other Names: Xadago

SUMMARY:
Patients suffering of Parkinson's Disease will be treated with 50 mg/day of Safinamide per os for 2 weeks (escalation phase). Then, safinamide will be increased up to 100 mg/day and, if tolerated, the treatment will be taken for 10 more weeks (maintenance phase). Total treatment 12 weeks.

DETAILED DESCRIPTION:
Adult patients affected by PD and suffering from motor fluctuations will be screened for participation.

If the inclusion and exclusion criteria are met, the participant will enter in the baseline assessment phase and undergo 1 night baseline PSG and 1 week baseline actigraphy. The patient will then start the treatment with 50 mg/day of Safinamide per os for 2 weeks (escalation phase). Then, safinamide will be increased up to 100 mg/day and, if tolerated, the treatment will last for 10 weeks (maintenance phase). At week 12 (end of treatment), the questionnaires, actigraphy and PSG will be repeated. A safety follow-up visit is scheduled 4 weeks after study treatment completion.

The treatment will be continued thereafter in all patients if medically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Fluctuating idiopathic PD patients according to UK Brain bank Criteria
* Hoehn and Year II to IV under treatment
* Sleep disturbance with a Pittsburgh Sleep Quality Index (PSQI) > 5
* Treatment with L-DOPA, alone or with other dopaminergic drugs, at a stable dose since at least 28 days prior to inclusion
* Treatment with all substances potentially acting on sleep and mood must be constant since at least 28 days prior to inclusion
* Written informed consent
* Willingness and ability to participate in the trial

Exclusion Criteria:

* Off label use of safinamide
* Early PD or absence of PD fluctuations
* Concomitant treatment with other MAO-B inhibitors (wash-out period: at least 14 days)
* Atypical Parkinsonism
* Severe known sleep-related breathing disorders with any specific treatment or severe known sleep-related breathing disorders (apnoea-hypopnea index score >30/h) with or without a specific treatment
* Dementia (MoCA < 26)
* Severe depression (BDI-II ≥ 29)
* Other severe psychiatric symptoms such as active psychosis or major hallucinations
* Any previous or concomitant severe medical conditions or clinical laboratory abnormality which, in the clinical judgement of the Investigators, does not allow patients' participation into the study
* Moderate or severe hepatic impairment, any type of retinopathy and/or any pathology that is deemed to be a contraindication according to safinamide's SmPC
* Any concomitant treatment not allowed or contraindicated in the safinamide SmPC
* Women who are pregnant or breast feeding
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Effect of safinamide on overall sleep quality | 12 weeks
  To measure the change in PDSS-2 (Parkinson's Disease Sleep Scale Version 2) score and the changes in sleep maintenance (=total sleep time/partial sleep time) and sleep efficiency (=total sleep time/ time in bed) scores measured by polysomnography (PSG). PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance). Scores > 18 are considered as relevant sleep disturbances.

SECONDARY OUTCOMES:
Effect of safinamide on objective PSG sleep characterization | 12 weeks
  To determine neurophysiological sleep parameters from PSG recording
Effect of safinamide on subjective sleep quality and sleepiness | 12 weeks
  To measure the change in subjective sleep quality as measured by PDSS-2 subscores and by the electronic diary "Sleep Fit app", and in daytime sleepiness as measured by ESS (Epworth sleepiness scale) score. PDSS-2 total score ranges from 0 (no disturbance) to 60 (maximum nocturnal disturbance). Scores > 18 are considered as relevant sleep disturbances. ESS score ranges from 0 to 24. Scores > 10 suggest relevant daytime sleepiness.
Effect of safinamide on objective motor activity | 12 weeks
  To determine the change in motor activity as measured by a specific objective measure of bradykinesia (FitTest) in the electronic diary "Sleep Fit app".
Effect of safinamide on subjective motor activity | 12 weeks
  To measure the change in motor activity as measured by UPDRS (Unified Parkinson's Disease Rating Scale). Higher UPDRS score indicates more severe impairment of non-motor and motor activities.
Effect of safinamide on objective sleep parameters and motor symptoms | 12 weeks
  To measure the change in sleep parameters and motor activity during the day and the night as measured by actigraphy.
Effect of safinamide on non-motor symptoms | 12 weeks
  To measure the change in depressive symptoms as measured by (BDI-II) Beck Depression Inventory and SAS (Starkstein Apathy Scale). Total BDI-II score ranges from 0 to 63 with higher total score indicating more severe depressive symptoms. Total SAS score ranges from 0 to 42 with higher scores indicating more severe apathy.
Effect of safinamide on quality of life | 12 weeks
  To measure the change in quality of life as measured by PDQ-39 (Parkinson's Disease Questionnaire-39). PDQ-39 is scored on a scale of 0 to 100, with lower scores indicating better health and high scores more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Neurocenter of Southern Switzerland - Ente Ospedaliero Cantonale (EOC), Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided